CLINICAL TRIAL: NCT00149071
Title: Treatment of Therapy-Resistant Major Depression With Transcranial Stimulation rTMS in Combination With Escitalopram
Brief Title: Transcranial Magnetic Stimulation (rTMS) Accelerates the Response to Escitalopram in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Medicon Valley Academy (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1,2
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Major Depression
Keywords: Transcranial magnetic stimulation (TMS); Major depression; treatment resistant major depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): rTMS
  Interventions: Device: rTMS; Device: TMS
- B (Sham Comparator): sham rTMS
  Interventions: Device: TMS; Device: rTMS

INTERVENTIONS:
Device: rTMS — 15 treatments of rTMS active with a duration of 30 minutes each
  Arms: A
Device: TMS — Transcraniel Magnetic Stimulation active and sham
Device: rTMS — active Transcranial Magnetic Stimulation
Device: rTMS — daily for three weeks

SUMMARY:
A doubleblind randomised trial with active versus sham rTMS in combination with escitalopram in patients with prior treatment resistant depression in an acute 12 weeks trial with subsequent 24 weeks study phase with active versus placebo citalopram

DETAILED DESCRIPTION:
In this study we aimed at investigating to what degree rTMS applied over the left dorsolateral cortex relieves depressive symptoms when the treament is combined with antidepressive medication. The study will also be able to supply knowledge on how long any possible effect of the rTMS treatment lasts.

In the first 12 weeks of the trial participants are randomised to either rTMS combined with escitalopram or sham rTMS combined with escitalopram. rTMS is given daily for the first 3 weeks.

The next phase is a relapse prevention study where the responders from the initial phase are randomised to either active or placebo escitalopram for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Major depression Hamilton score above 18
* Age 18 to 75

Exclusion Criteria:

* Pregnancy og breastfeeding
* Mental retardation and organic brain disease
* Alcohol and substance abuse
* Metal implants in brain, pacemakers and other electronic implants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
depression scores | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Line G Bretlau, MD, Principal Investigator — Psychiatric research Unit, Hilleroed Hospital, Denmark
Locations (1):
- Psychiatric research unit, Hilleroed Hospital,, Hillerød, Denmark